CLINICAL TRIAL: NCT01015950
Title: Randomized, Community-Based Effectiveness Trial of Selected Dietary Strategies for the Management of Young Malian Children With Moderate Acute Malnutrition (MAM) in the Context of the National Community Management of Acute Malnutrition
Brief Title: Management of Children With Moderate Acute Malnutrition in Mali
Acronym: Mali-MMAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: University of Bamako (Other); University of California, Davis (Other); UNICEF (Other); United Nations World Food Programme (WFP) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200917501-1, 200917501-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Moderate Acute Malnutrition (MAM)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pumpy'Sup (Experimental): Lipid-based nutrient supplement
  Interventions: Dietary Supplement: Plumpy'Sup
- SCSB (Experimental): Processed, fortified, cereal-based food blend (SCSB for malnourished children)
  Interventions: Dietary Supplement: SCSB
- Misola (Experimental): Locally processed, fortified food blend (Misola)
  Interventions: Dietary Supplement: Misola
- Local food supplement (Active Comparator): Local foods (millet flour, cowpea flour, sugar, oil) and a multiple micronutrient powder ("Mix-Me") are provided to simulate the currently recommended enhanced home-prepared rehabilitation food mixture ("farines enrchies") according to the national Mali CMAM protocol.
  Interventions: Dietary Supplement: Local food supplement

INTERVENTIONS:
Dietary Supplement: Plumpy'Sup — Lipid-based (vegetable oil, peanut paste, soy protein-containing) fortified nutrient supplement to provide 500 kcal/d
  Other Names: Plumpy'Sup, Supplementary Plumpy, Nutriset, France
  Arms: Pumpy'Sup
Dietary Supplement: Local food supplement — Local foods (millet flour, cowpea flour, sugar, vegetable oil) and a multiple micronutrient powder ("Mix Me") are provide, according to the national Mali CMAM protocol when special processed foods are not available.
  Arms: Local food supplement
Dietary Supplement: Misola — Locally produced, millet-soy-peanut-based fortified complementary food (Misola)
  Other Names: Misola, Mali
  Arms: Misola
Dietary Supplement: SCSB — Processed, fortified, corn-soy-milk-based food blend (SCSB for malnourished children, to be supplied by the World Food Program) to provide an additional 500 kcal/day
  Other Names: World Food Program
  Arms: SCSB

SUMMARY:
The objectives of the study are to assess the impact of different dietary strategies for the management of children with MAM on: the children's continued participation in the nutritional rehabilitation program and their physical growth, recovery from MAM, and change in micronutrient status and body composition. The specific dietary regimens that will be compared are: 1) a ready-to-use, lipid-based supplementary food (Plumpy'Sup, Nutriset, Inc.), providing ~500 kcal/d for 12 weeks; 2) specially formulated CSB for malnourished children, providing ~ 500 kcal/d for 12 weeks; 3) Misola, a locally produced, micronutrient-fortified, cereal-legume blend, providing ~500 kcal/d for 12 weeks; or 4) packaged, home available foods (millet and cowpea flour, sugar, vegetable oil) and a multiple micronutrient powder ("Mix Me") for 12 weeks, as is currently recommended by the national CMAM protocol when special foods are not available.

ELIGIBILITY:
Inclusion Criteria:

* age from 6 to 35 months,
* MUAC <12.5 cm and >11.0 cm, and weight-for-length (WLZ) Z-score > -3.0 (WHO standard, 2006); or WLZ <-2.0 and >-3.0 and MUAC >11.0 cm
* absence of bi-pedal edema
* absence of current diseases requiring inpatient care
* expected availability during the period of the study
* residency within the study communities
* acceptance of home visitors, and
* written consent of a parent or guardian

Exclusion Criteria:

* age <6 months or >36 months
* MUAC >12.5 cm and WLZ >-2.0; or MUAC <11.0 cm; or WLZ <-3.0
* presence of bi-pedal edema,
* severe anemia (defined as hemoglobin <50 g/L),
* other acute illnesses requiring inpatient treatment,
* congenital abnormalities or underlying chronic diseases, including known HIV . infection, that may affect growth or risk of infection
* history of allergy towards peanuts or previous serious allergic reaction to . any substance, requiring emergency medical care
* concurrent participation in any other clinical trial

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1260 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight gain | 3 months
Continuation in treatment | 3 months

SECONDARY OUTCOMES:
Micronutrient status | 3 months
Body composition | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — Helen Keller International
Locations (1):
- Helen Keller International, Bamako, Mali

REFERENCES:
- [Derived] Isanaka S, Barnhart DA, McDonald CM, Ackatia-Armah RS, Kupka R, Doumbia S, Brown KH, Menzies NA. Cost-effectiveness of community-based screening and treatment of moderate acute malnutrition in Mali. BMJ Glob Health. 2019 Apr 28;4(2):e001227. doi: 10.1136/bmjgh-2018-001227. eCollection 2019. PMID 31139441
- [Derived] McDonald CM, Ackatia-Armah RS, Doumbia S, Kupka R, Duggan CP, Brown KH. Percent Fat Mass Increases with Recovery, But Does Not Vary According to Dietary Therapy in Young Malian Children Treated for Moderate Acute Malnutrition. J Nutr. 2019 Jun 1;149(6):1089-1096. doi: 10.1093/jn/nxz037. PMID 30968123
- [Derived] Ackatia-Armah RS, McDonald CM, Doumbia S, Erhardt JG, Hamer DH, Brown KH. Malian children with moderate acute malnutrition who are treated with lipid-based dietary supplements have greater weight gains and recovery rates than those treated with locally produced cereal-legume products: a community-based, cluster-randomized trial. Am J Clin Nutr. 2015 Mar;101(3):632-45. doi: 10.3945/ajcn.113.069807. Epub 2015 Jan 7. PMID 25733649